CLINICAL TRIAL: NCT05643222
Title: The Performance of Red Tinted Contact Lenses of Various Tones on Colour Deficient Subjects: A Pilot Study
Brief Title: Performance of Red Tinted Contact Lenses on Colour Defects
Acronym: CL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: UKM PPI/111/8/JEP-2021-145
Record Dates: First submitted 2022-11-21; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Color Vision Defects; Color Blindness
Keywords: Anomalous Trichromats; Color Vision Defect; Contact Lenses
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Intervention Model Description: 6 colour defect subjects eye were inserted with 4 different types of red tinted contact lenses at different times and then tested with Ishihara Test and 100 Hue Test to obtain the score values. This was done only on one non dominant eye of subject.
Who Masked: Outcomes Assessor
Masking Description: Only the principal investigator knows the identity of each of the lenses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TES and performance assessment with Type A Red Tint Lens (Active Comparator): 6 subjects will be inserted with the Type A red Tint Lenses. Only the non dominant eye will be inserted. The comparison is made before and after wearing the CL.
  Interventions: Device: red tint contact lenses
- TES and performance assessment with Type B Red Tint Lens (Active Comparator): 6 subjects will be inserted with the Type B red Tint Lenses. Only the non dominant eye will be inserted. The comparison is made before and after wearing the CL.
  Interventions: Device: red tint contact lenses
- TES and performance assessment with Type C Red Tint Lens (Active Comparator): 6 subjects will be inserted with the Type C red Tint Lenses. Only the non dominant eye will be inserted. The comparison is made before and after wearing the CL.
  Interventions: Device: red tint contact lenses
- TES and performance assessment with Type D Red Tint Lens (Active Comparator): 6 subjects will be inserted with the Type D red Tint Lenses. Only the non dominant eye will be inserted. The comparison is made before and after wearing the CL.
  Interventions: Device: red tint contact lenses

INTERVENTIONS:
Device: red tint contact lenses — to compare the performance of these lenses.
  Other Names: IGEL Red tint lens type1; IGEL Red tint lens type 2; OCULUS Red tint lens; MAXVUE Red tint lens

SUMMARY:
This study aimed to relate and compare the performance of 4 types of red-tinted contact lenses (CL) with the Total Error Score (TES) from the Farnsworth-Munsell 100 Hue test on colour deficient subjects. Only 6 subject with colour vision defect was tested in this study.

DETAILED DESCRIPTION:
Six congenital CVD subjects were recruited. After colour vision screening using Ishihara plate, the Farnsworth-Munsell 100 Hue test was carried out to determine the type and severity of colour vision deficiency. Four types of red-tinted CL (Type A, B, C and D) were used. The performance of each of these lenses was determined through the comparison of error scores in the Ishihara test before and after wearing tinted contact lens on only the non-dominant eye. Then, the transmittance of each tinted CL was determined using a spectrophotometer. All these lenses were fitted on the subjects in one day where the subjects were given a 30-minute break for each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-40 years
* all sex
* color defect diagnosed with Ishihara Test
* no contraindication in contact lens wear

Exclusion Criteria:

* have ocular and systemic diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
The lens which gives the best result in TES value | 30 minutes after lens adaptation. Lens is removed immediately after the assessment is completed.
  The highest TES value scored showed higher performance in colour vision. TES is an automated, generated value that calculates the number of tiles placed incorrectly and scales the value for uniform analysis. Average TES scores range from thirty to forty in series tests; while scores exceeding seventy can point to a marker for color blindness. Lower scores are intended to point to significantly increased color vision accuracy, as the TES score is directly correlated to the number of tiles incorrectly identified
The lens which gives the best performance in ES value | 30 minutes after lens adaptation. Lens is removed immediately after the assessment is completed
  The highest score achieved using Ishihara Test indicates the best red tint lens. The current passing score is 12 correct of 14 red/green test plates (not including the demonstration plate). Research has shown that scores below twelve indicate color vision deficiency, and twelve or more correct indicate normal color vision, with 97% sensitivity and 100% specificity

CONTACTS AND LOCATIONS:
Overall Officials: Haliza Abdul Mutalib, PhD, Principal Investigator — UKM
Locations (1):
- Optometry Clinic, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
only the executive summary of all data analysis published by journals will be made available. IPD will be shared only when requested.

REFERENCES:
- [Background] Cole BL, Lian KY, Lakkis C. Using clinical tests of colour vision to predict the ability of colour vision deficient patients to name surface colours. Ophthalmic Physiol Opt. 2007 Jul;27(4):381-8. doi: 10.1111/j.1475-1313.2007.00493.x. PMID 17584289

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Informed Consent (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT05643222/Prot_SAP_ICF_000.pdf
  • Study Protocol: Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT05643222/Prot_001.pdf